CLINICAL TRIAL: NCT02918864
Title: Integrated Oxytocin and Nonverbal, Emotion Recognition, and Theory of Mind Training for Children With Autism Spectrum Disorder
Brief Title: Oxytocin and Social Cognitive Skills Groups
Acronym: ION-ASD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: University of Illinois at Chicago (Other); University of Chicago (Other); Northwestern University (Other); Eotvos Lorand University (Other)
Responsible Party: Principal Investigator, Latha Soorya, Assistant Professor of Psychiatry, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14062403
Record Dates: First submitted 2016-09-09; First posted 2016-09-29 (Estimated); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Oxytocin; Social Skills; Social cognitive skills; Cognitive Behavioral Intervention; Combination treatment; Syntocinon; NETT (Nonverbal communication, Emotion recognition, Theory of mind Training); emotion recognition; theory of mind
MeSH Terms: conditions — Autism Spectrum Disorder; Social Skills; Nonverbal Communication | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ION-ASD (Experimental): ION-ASD integrates targeted dosing of intranasal oxytocin and social cognitive skills group training curriculum, Seaver-NETT (Nonverbal communication, Emotion recognition, Theory of mind Training).
  Interventions: Drug: Oxytocin; Behavioral: Social Cognitive Skills Training
- Facilitated Play (Active Comparator): The active comparison condition is a facilitated play therapy group.
  Interventions: Behavioral: Facilitated Play Therapy

INTERVENTIONS:
Drug: Oxytocin — This is an integrated pharmacological-behavioral intervention targeting social cognitive skills for school-aged children with ASD. Four doses of intranasal oxytocin (24 IUs/dose) will be delivered each week before weekly homework and group therapy sessions.
  Other Names: Syntocinon
  Arms: ION-ASD
Behavioral: Social Cognitive Skills Training — Social cognitive skills training utilize cognitive behavioral strategies such as problem identification, affective education, performance feedback, and weekly homework activities to target impairments in nonverbal synchrony, emotional expression, and interpretation of intent. The NETT curriculum is manualized and anchored in CBI strategies, such as problem identification, affective education, performance feedback, and weekly homework activities. Parent education sessions run concurrently with child groups to help facilitate generalization.
  Other Names: NETT
  Arms: ION-ASD
Behavioral: Facilitated Play Therapy — The facilitated play therapy group is a manualized treatment designed to tailor play to the interests and abilities of group members. Therapists use general therapeutics strategies such as reflective functioning statements to foster communication with therapists as well as between peers. Standard educational practices for children with ASD such as visual supports, schedules, and short-directed statements are also used. The concurrent parent group is supportive in nature.
  Arms: Facilitated Play

SUMMARY:
The purpose of this study is to evaluate the feasibility, safety, and preliminary efficacy of integrating targeted dosing of intranasal oxytocin with a social cognitive skills group therapy for school-aged children with autism spectrum disorder (ASD).

DETAILED DESCRIPTION:
The study is a proof-of-concept, combination intervention designed to address individual treatment targets presumed to influence social learning in school-aged children with autism spectrum disorder (ASD). This proposal builds upon prior research on an empirically supported social cognitive skills training curriculum, NETT (Nonverbal communication, Emotion recognition, and Theory of mind Training). NETT is a cognitive-behavioral intervention (CBI) for nonverbal communication, emotion recognition, and theory of mind deficits in youth with ASD. In this two-phase, 3 year, single-blind, contact controlled study, school-aged children with ASD (n=60) will be randomized into a 12-session, parallel group design of Integrated Oxytocin and NETT (ION) or a control social group condition (facilitated play). The study aims to evaluate the safety, tolerability, and efficacy of integrating the neuropeptide, oxytocin (OXT), with the social cognitive curriculum, as well as to identify targets of change and pre-treatment factors predictive of response to ION-ASD. Maintenance of treatment effects will also be assessed 1 month and 3 months post-treatment.

ELIGIBILITY:
Inclusion Criteria

1. Male or female outpatients, 8-11 years of age inclusive
2. Meet Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) for Autism Spectrum Disorder. DSM-V criteria will be established by a clinician with expertise with individuals with ASD. Best estimate Diagnosis will be reached using DSM-5 criteria, the Autism Diagnostic Observation Schedule (ADOS-2) and the Autism Diagnostic Interview (ADI-R), or Autism Screening Interview.
3. Mean score of 9 or less on mentalizing items of Strange Stories Test (Highest possible score = 12, items 21-25, 27).
4. Have a Clinician's Global Impression-Severity (CGI-S) score ≥ 4 (moderately ill) at Baseline.
5. Verbal and performance scale intelligence quotient (IQ) ≥ 80 (both subtests of the Wechsler Intelligence Scale for Children-V (WISC-V) ≥ 70).
6. If already receiving stable concomitant medications, have continuous participation during the preceding 30 days prior to Screening, and not electively initiate new or modify ongoing medications for the duration of the study. For serotonergic agents, 6 months on a stable dose is required.
7. If already receiving stable non-pharmacologic educational, behavioral, and/or dietary interventions, have continuous participation during the preceding 3 months prior to Screening, and not electively initiate new or modify ongoing interventions for the duration of the study.
8. Have normal physical examination and laboratory test results at Screening. If abnormal, the finding(s) must be deemed not clinically significant by the Treating Clinician.
9. Ability to speak and understand English sufficiently to allow for the completion of all study assessments.
10. Ability to obtain written assent from the participant as well as written informed consent from their parent(s)/legal guardian.

Exclusion Criteria

1. Patients born prior to 35 weeks gestational age.
2. Patients with a primary psychiatric diagnosis other than ASD.
3. Patients with a medical history of neurological disease, including, but not limited to, epilepsy/seizure disorder (except simple febrile seizures), movement disorder, tuberous sclerosis, fragile X, and any other known genetic syndromes, or known abnormal brain MRI/structural lesion.
4. Pregnant female patients, sexually active female patients on hormonal birth control and sexually active females who do not use at least two types of non-hormonal birth control.
5. Patients with evidence or history of malignancy or any significant hematological, endocrine, cardiovascular (including any rhythm disorder), respiratory, renal, hepatic, or gastrointestinal disease.
6. Patients with one or more of the following: hemophilia (bleeding problems, recent nose and brain injuries), abnormal blood pressure (hypotension or hypertension), drug abuse, immunity disorder or severe depression.
7. Patients who are currently taking oxytocin (OXT) or have taken intranasal oxytocin (IN-OXT) in the past with no response.
8. Patients who have an Aberrant Behavior Checklist (ABC) Irritability subscale score > 19 at screening
9. Patients with sensitivity to OXT or any components of its formulation.
10. Patients unable to tolerate venipuncture procedures for blood sampling.
11. Patients in foster care for whom the state is defined as a legal guardian.
12. If they have an arrhythmia present on ECG, that upon consultation with a cardiologist, is deemed to be clinically significant.
13. Patients with any of the following clinical lab results

    1. Alanine transaminase (ALT) or aspartate transaminase (AST) levels of ≥ 5 times the upper limit of normal, or if clinical jaundice occurs
    2. Sodium levels of > 152 mmol/L or < 128 mmol/L
    3. Potassium levels of > 6 mmol/L in a non-hemolyzed sample
    4. Glucose levels of > 11 mmol/L or < 2.8 mmol/L
    5. Hemoglobin levels of < 100 g/L
    6. Blood urea nitrogen (BUN) levels of > 100 mmol/L
    7. Creatinine levels of > 100 µmol/L
    8. Osmolality levels of > 330 mmol/kg

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Latha Soorya, PhD, BCBA, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be submitted to the National Database for Autism Research (NDAR), a computer system run by the National Institutes of Health that allows researchers studying autism to collect and share information. Data will be shared with study collaborators as well.

REFERENCES:
- [Background] Soorya LV, Siper PM, Beck T, Soffes S, Halpern D, Gorenstein M, Kolevzon A, Buxbaum J, Wang AT. Randomized comparative trial of a social cognitive skills group for children with autism spectrum disorder. J Am Acad Child Adolesc Psychiatry. 2015 Mar;54(3):208-216.e1. doi: 10.1016/j.jaac.2014.12.005. Epub 2014 Dec 20. PMID 25721186

RESULTS

PARTICIPANT FLOW:
Groups:
- ION-ASD: ION-ASD integrates targeted dosing of intranasal oxytocin and social cognitive skills group training curriculum, Seaver-NETT (Nonverbal communication, Emotion recognition, Theory of mind Training).
  Oxytocin: This is an integrated pharmacological-behavioral intervention targeting social cognitive skills for school-aged children with ASD. Four doses of intranasal oxytocin (24 IUs/dose) will be delivered each week before weekly homework and group therapy sessions.
  Social Cognitive Skills Training: Social cognitive skills training utilize cognitive behavioral strategies such as problem identification, affective education, performance feedback, and weekly homework activities to target impairments in nonverbal synchrony, emotional expression, and interpretation of intent. The NETT curriculum is manualized and anchored in cognitive behavioral intervention (CBI) strategies, such as problem identification, affective education, performance feedback, and weekly homework activities. Parent education sessions run concurrently with child groups to help facilitate generalization.
Period: Overall Study
Arm/Group | ION-ASD | Facilitated Play
Started | 20 | 20
Endpoint (Week 12) | 19 | 19
1-month Follow-up (Week 16) | 17 | 18
3-month Follow-up (Week 24) | 16 | 17
Completed | 16 | 17
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ION-ASD | Facilitated Play | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.30 (1.13) | 9.20 (1.11) | 9.25 (1.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 19 | 18 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 7 | 10 | 17
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 4 | 3 | 7
CCC-2 Nonverbal Communication [Mean (Standard Deviation); unit: units on a scale] — The Children's Communication Checklist-2 (CCC-2) Nonverbal subscale contains 7 items scored on a 4-point scale (0/less than once a week to 3/every day) for a total range of 0-21; higher total scores reflect greater impairment. Items estimate children's nonverbal communication skills (e.g., eye contact, social distance recognizing other's emotions) and are dispersed in a 70-item parent questionnaire intended for children 4-16-years-old.
  units on a scale | 8.80 (4.28) | 8.75 (3.26) | 8.77 (3.75)
CCC-2 Social Relations [Mean (Standard Deviation); unit: units on a scale] — The Children's Communication Checklist-2 (CCC-2) Social Relations subscale contains 7 items scored on a 4-point scale (0/less than once a week to 3/every day) for a total range of 0-21; higher total scores reflect greater impairment. Items estimate children's social competence (e.g., comfort around others, sensitivity to and interest in others) and are dispersed in a 70-item parent questionnaire intended for children 4-16-years-old.
  units on a scale | 8.30 (3.80) | 7.60 (2.33) | 7.95 (3.13)
Griffith Empathy Measure [Mean (Standard Deviation); unit: units on a scale] — The Griffith Empathy Measure (GEM) is a brief parent report survey adapted from an adult empathy measure intended to capture cognitive (i.e., identifying another's situation and taking their perspective) and affective (i.e., responding according to the other's perspective rather than one's own) empathy skills in pre- and through adolescence. Total scores range from -92 to 92, the sum of 23 items scored on a 9-point scale (-4/strongly disagree to 4/strongly agree), with lower total scores reflecting greater impairment.
  units on a scale | 12.65 (19.02) | 22.05 (20.20) | 17.35 (19.94)
RMET, % correct [Mean (Standard Deviation); unit: percentage of correct items] — Reading the Mind in the Eyes Test (RMET) % correct out of items administered (maximum 28), participant task
  percentage of correct items | 63.57 (14.96) | 58.93 (19.82) | 61.25 (17.49)
DANVA2, % correct [Mean (Standard Deviation); unit: percentage of correct items] — Diagnostic Analysis of Nonverbal Accuracy-2 (DANVA2) % correct out of items administered (maximum 96), participant task
  percentage of correct items | 65.23 (16.32) | 65.86 (11.92) | 65.55 (14.11)
Verbal IQ [Mean (Standard Deviation); unit: units on a scale] — Wechsler Abbreviated Scale of Intelligence, 2nd ed (WASI-II) and Wechsler Intelligence Scale for Children, 4th ed (WISC-IV) are clinician administered intelligence tests. Both tests provide a full scale, non-verbal and verbal intelligence quotient (IQ). Verbal IQ is estimated using the Verbal Comprehension Index (VCI). The WASI-II Vocabulary and Similarities subtests form the VCI. The WISC-IV Vocabulary, Similarity, and Comprehension subtests form the VCI. VCI provides an estimated verbal IQ ranging from 40-160, mean of 100 (standard deviation of 15); higher scores indicate better performance. Population: Data was missing for one participant's VIQ
  units on a scale
    number analyzed (Participants) | 20 | 19 | 39
    (all) | 96.30 (18.16) | 99.84 (18.24) | 98.03 (18.05)
ADHD CASI-5 T-score [Mean (Standard Deviation); unit: T-score] — The Attention Deficit Hyperactivity Disorder (ADHD) combined subscale from the Child & Adolescent Symptom Inventory-5 (CASI-5) measures the frequency of ADHD symptoms in children ages 5-18-years-old. Parents rate the frequency of 18 behavioral items on a 173-item form from 0/never to 3/very often. Items scores are totaled, and raw total subscale scores are converted into ADHD symptom severity T-scores for youth (5-12 yo) by sex. T-scores have a normative mean of 50 (SD=10) with severity categorized as 50-59/low, 60-69/moderate, 70 and above/high indicating clinical impairment.
  T-score | 69.80 (14.24) | 69.70 (9.56) | 69.75 (11.97)
Social Responsiveness Scale-2 (SRS-2) [Mean (Standard Deviation); unit: T-score] — The SRS-2 is a caregiver reported measure of social behavior in the general population (3-18 yo) used to assess social functioning. The SRS-2 contains 65 items rated on a 4-point scale (1/not true to 4/almost always true). Scores are recoded 0-3 and totaled for a raw score. Raw scores convert to T-scores using age and sex. T-scores have a population mean of 50 with a standard deviation of 10. T-scores 60-65 indicate mild social impairment, 66-75 moderate deficits, and above 76 severe deficits strongly associated with autism. Higher SRS-2 T-scores indicate greater severity of social impairment.
  T-score | 71.25 (11.09) | 69.50 (8.43) | 70.38 (9.76)
Caregiver Strain Questionnaire-Global Strain (CGSQ) [Mean (Standard Deviation); unit: units on a scale] — The CGSQ was used to assess quality of life. The CGSQ is a parent-rated questionnaire designed for parents of children and adolescents with emotional and behavioral disorders. It includes 21 items rated on a 5-point problem scale (1 = not at all to 5 = very much) rating subjective internal, subjective external, and objective strain. A global measure of strain can be calculated by averaging the scores together. Higher CGSQ scores indicate greater strain.
  units on a scale | 2.52 (0.79) | 2.24 (0.51) | 2.38 (0.67)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Social Behavior Impairment (SBI) Composite
Description: The change from baseline in SBI is represented by the slope of each group. The primary outcome is the difference between groups in this rate of change or the group*time interaction. SBI is a composite score based on Soorya et al. (2015) which identified measures that comprise this metric. Scores from the Children's Communication Checklist-2 (CCC-2) Social Relations and Nonverbal Communication subscales and the Griffith Empathy Measure (GEM) were standardized as z-scores using the sample means and standard deviations at baseline. CCC-2 subscale scores and reversed GEM total scores were used so higher z-scores reflect more impairment across measures. The SBI outcome was subsequently derived by averaging the z-scores. At baseline, the sample average SBI z-score equals 0; higher individual scores indicate relatively more impairment in social behavior skills. Larger, negative slopes represent improvement.
Time Frame: Baseline and Week 12 (Endpoint)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: z-score
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
z-score
  Estimated mean (baseline) | 0.12 (0.14) | -0.14 (0.14)
  Estimated mean (week 12) | -0.26 (0.14) | -0.16 (0.14)
Statistical Analysis 1: Comparison: ION-ASD vs Facilitated Play; Ho=No significant interaction of Group*Time; Test type: Superiority; p = 0.037, Mixed Models Analysis — p-value reported for Group*Time, primary comparison in linear mixed effects model (SB=Group+Time+Group*Time+ADHD+ γ + ε; ADHD, CASI T-score significant covariate), not adjusted for multiple tests (with different time points); Beta Coefficient = -.22

2. Primary Outcome: Rate of Change From Baseline in Social Behavior Impairment (SBI) Composite
Description: as for outcome 1
Time Frame: Baseline and Week 12 (Endpoint)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: scores/week
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
scores/week | -0.03 (0.01) | 0.00 (0.01)

3. Primary Outcome: Change From Baseline in Social Behavior Impairment (SBI) Composite
Description: as for outcome 1
Time Frame: Baseline and Week 16 (1-month follow-up)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: z-score
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
z-score
  Estimated mean (baseline) | 0.11 (0.13) | -0.14 (0.14)
  Estimated mean (week 16) | -0.29 (0.14) | -0.14 (0.14)
Statistical Analysis 1: Comparison: ION-ASD vs Facilitated Play; Ho=No significant interaction of Group*Time; Test type: Superiority; p = 0.016, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Beta Coefficient = -.23

4. Primary Outcome: Rate of Change From Baseline in Social Behavior Impairment (SBI) Composite
Description: as for outcome 1
Time Frame: Baseline and Week 16 (1-month follow-up)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: scores/week
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
scores/week | -0.03 (0.01) | 0.00 (0.01)

5. Primary Outcome: Change From Baseline in Social Behavior Impairment (SBI) Composite
Description: as for outcome 1
Time Frame: Baseline and Week 24 (3-month follow-up)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: z-score
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
z-score
  Estimated mean (baseline) | 0.04 (0.14) | -0.16 (0.14)
  Estimated mean (week 24) | -0.21 (0.15) | -0.08 (0.15)
Statistical Analysis 1: Comparison: ION-ASD vs Facilitated Play; Ho=No significant interaction of Group*Time; Test type: Superiority; p = 0.061, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Beta Coefficient = -.16

6. Primary Outcome: Rate of Change From Baseline in Social Behavior Impairment (SBI) Composite
Description: as for outcome 1
Time Frame: Baseline and Week 24 (3-month follow-up)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: scores/week
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
scores/week | -0.01 (0.01) | 0.00 (0.00)

7. Primary Outcome: Change From Baseline in Social Cognition (SC) Composite
Description: The change from baseline in SC is represented by the slope of each group. The primary outcome is the difference between groups in this rate of change or the group*time interaction. SC is a composite score, including the Reading the Mind in the Eyes Test (RMET) and the Diagnostic Analysis of Nonverbal Accuracy-2 (DANVA2), based on Soorya et al. (2015). RMET has 28 items rated correct/incorrect (total 0-28). DANVA2 contains 4 sets of 24 items rated correct/incorrect (total 0-96). Percent correct was calculated for each measure given the difference in denominators and to allow for administrative omissions. Percentages were standardized as z-scores using the sample means and standard deviations at baseline. The SC outcome was subsequently derived by averaging the z-scores. At baseline, the sample average SC z-score equals 0; higher individual scores reflect stronger skills on social cognitive tasks compared to lower scores. Larger, positive slopes indicate skill improvement.
Time Frame: Baseline and Week 12 (Endpoint)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: z-score
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
z-score
  Estimated mean (baseline) | 0.06 (0.18) | -0.08 (0.18)
  Estimated mean (week 12) | 0.37 (0.18) | 0.16 (0.19)
Statistical Analysis 1: Comparison: ION-ASD vs Facilitated Play; Ho=No significant interaction of Group*Time; Test type: Superiority; p = 0.674, Mixed Models Analysis — p-value reported for Group*Time, primary comparison in linear mixed effects model (SC=Group+Time+Group*Time+Group*VIQ+ γ + ε; VIQ, verbal intelligence quotient (VIQ) significant moderator), not adjusted for multiple tests (with different time points); Beta Coefficient = 0.03

8. Primary Outcome: Rate of Change From Baseline in Social Cognition (SC) Composite
Description: as for outcome 7
Time Frame: Baseline and Week 12 (Endpoint)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: scores/week
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
scores/week | 0.03 (0.01) | 0.02 (0.01)

9. Primary Outcome: Change From Baseline in Social Cognition (SC) Composite
Description: as for outcome 7
Time Frame: Baseline and Week 16 (1-month follow-up)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: z-score
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
z-score
  Estimated mean (baseline) | 0.06 (0.18) | -0.08 (0.18)
  Estimated mean (week 16) | 0.57 (0.17) | 0.25 (0.18)
Statistical Analysis 1: Comparison: ION-ASD vs Facilitated Play; Ho=No significant interaction of Group*Time; Test type: Superiority; p = 0.191, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Beta Coefficient = 0.09

10. Primary Outcome: Rate of Change From Baseline in Social Cognition (SC) Composite
Description: as for outcome 7
Time Frame: Baseline and Week 16 (1-month follow-up)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: scores/week
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
scores/week | 0.03 (0.01) | 0.02 (0.01)

11. Primary Outcome: Change From Baseline in Social Cognition (SC) Composite
Description: as for outcome 7
Time Frame: Baseline and Week 24 (3-month follow-up)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: z-score
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
z-score
  Estimated mean (baseline) | 0.10 (0.17) | -0.08 (0.17)
  Estimated mean (week 24) | 0.63 (0.17) | 0.37 (0.17)
Statistical Analysis 1: Comparison: ION-ASD vs Facilitated Play; H0=No significant interaction of Group*Time; Test type: Superiority; p = 0.599, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Beta Coefficient = 0.04

12. Primary Outcome: Rate of Change From Baseline in Social Cognition (SC) Composite
Description: as for outcome 7
Time Frame: Baseline and Week 24 (3-month follow-up)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: scores/week
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
scores/week | 0.02 (0.00) | 0.02 (0.00)

13. Secondary Outcome: Number of Responder and Non-responder Participants Based on CGI-I Scores at Week 12 (Endpoint)
Description: Global Functioning will be assessed using the Clinical Global Impressions-Improvement (CGI-I) Scale. A study physician followed standard CGI protocols to evaluate global improvement at each time point based on all available sources of information (e.g., caregiver interviews, behavior rating forms). The CGI-I employs a 7-point scale with the lowest score, 1, indicating the best outcome and the highest score, 7, indicating the worst outcome. Participants receiving scores of 1 (very much improved) or 2 (much improved) were considered responders. Participants receiving scores of 5 (minimally worse), 6 (much worse), or 7 (very much worse) were considered non-responders; note, no participant received a score worse than 5 which was used as the cut-off for non-responders. Participants receiving scores of 3 (minimally improved) or 4 (no change) were considered to show no significant change and omitted from the analysis.
Time Frame: Week 12 (Endpoint)
Population: If participants were missing CGI-I ratings at week 12 (Facilitated Play: n=2), the rating from the last available visit (i.e., week 6) was used. Participants with scores of 3 or 4, indicating no significant change, were not included in the responder analyses (ION-ASD: n=12; Facilitated Play: n=12). One participant (Facilitated Play) had no data to carry forward. Additionally, two participants dropped out of the study (ION-ASD: n=1; Facilitated Play: n=1) and were excluded from the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 7 | 6
Participants
  Responder (scores 1-2) | 7 | 5
  Non-responder (score 5-7) | 0 | 1
Statistical Analysis 1: Comparison: ION-ASD vs Facilitated Play; Ho=Group and response are independent (responders="improved" scores of 1-2; non-responders="worsened" scores of 5-7 on the CGI-I) at week 12; Test type: Superiority; p = 0.462, Fisher Exact — 2-sided p-value; p-value reported not adjusted for multiple tests (with different time points)

14. Secondary Outcome: Number of Responder and Non-responder Participants Based on CGI-I Scores at Week 16 (1-month Follow-up)
Description: as for outcome 13
Time Frame: Week 16 (1-month follow-up)
Population: If participants were missing CGI-I ratings at week 16 (ION-ASD: n=1; Facilitated Play: n=5), the rating from the last available visit (i.e., 5 from week 12 and 1 from week 6) was used. Participants with scores of 3 or 4, indicating no significant change, were not included in the responder analyses (ION-ASD: n=10; Facilitated Play: n=12). Additionally, from baseline to week 16, five participants dropped out of the study (ION-ASD: n=3; Facilitated Play: n=2) and were excluded from the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 7 | 6
Participants
  Responder (score 1-2) | 4 | 4
  Non-responder (score 5-7) | 3 | 2
Statistical Analysis 1: Comparison: ION-ASD vs Facilitated Play; Ho=Group and response are independent (responders="improved" scores of 1-2; non-responders="worsened" scores of 5-7 on the CGI-I) at week 16; Test type: Superiority; p = 1.000, Fisher Exact — 2-sided p-value; p-value reported not adjusted for multiple tests (with different time points)

15. Secondary Outcome: Number of Responder and Non-responder Participants Based on CGI-I Scores at Week 24 (3-month Follow-up)
Description: Global Functioning will be assessed using the Clinical Global Impressions-Improvement (CGI-I) Scale. A study physician followed standard CGI protocols to evaluate global improvement at each time point based on all available sources of information (e.g., caregiver interviews, behavior rating forms). The CGI-I employs a 7-point scale with the lowest score, 1, indicating the best outcome and the highest score, 7, indicating the worst outcome. Participants receiving scores of 1 (very much improved) or 2 (much improved) were considered responders. Participants receiving scores of 5 (minimally worse), 6 (much worse), or 7 (very much worse) were considered non-responders; note, no participant received a score worse than 5 which was used as the cut-off for non-responders . Participants receiving scores of 3 (minimally improved) or 4 (no change) were considered to show no significant change and omitted from the analysis.
Time Frame: Week 24 (3-month follow-up)
Population: If participants were missing CGI-I ratings at week 24 (ION-ASD: n=2), the rating from the last available visit (i.e., week 16) was used. Participants with scores of 3 or 4, indicating no significant change, were not included in the responder analyses (ION-ASD: n=6; Facilitated Play: n=11). Additionally, from baseline to week 24, seven participants dropped out of the study (ION-ASD: n=4; Facilitated Play: n=3) and were therefore excluded from the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 10 | 6
Participants
  Responder (score 1-2) | 7 | 3
  Non-responder (score 5-7) | 3 | 3
Statistical Analysis 1: Comparison: ION-ASD vs Facilitated Play; Ho=Group and response are independent (responders="improved" scores of 1-2; non-responders="worsened" scores of 5-7 on the CGI-I) at week 24; Test type: Superiority; p = 0.607, Fisher Exact — 2-sided p-value; p-value reported not adjusted for multiple tests (with different time points)

16. Secondary Outcome: Change From Baseline in Social Functioning (SRS-2)
Description: The change from baseline in the Social Responsiveness Scale (SRS-2) is represented by the slope of each group. The primary outcome is the difference between groups in this rate of change or the group*time interaction. The SRS-2 is a caregiver reported measure of social behavior in the general population (3-18 yo) used to assess social functioning. The SRS-2 contains 65 items rated on a 4-point scale (1/not true to 4/almost always true). Scores are recoded 0-3 and totaled for a raw score. Raw scores are converted to T-scores based on age and sex. T-scores have a population mean of 50 with a standard deviation of 10. T-scores 60-65 indicate mild social impairment, 66-75 moderate deficits, and above 76 severe deficits strongly associated with autism. Higher SRS-2 T-scores indicate greater severity of social impairment. Larger, negative slopes reflect a greater reduction in severity.
Time Frame: Baseline and Week 12 (Endpoint)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
T-score
  Estimated mean (baseline) | 70.83 (2.16) | 69.50 (2.22)
  Estimated mean (week 12) | 66.48 (2.38) | 68.79 (2.39)
Statistical Analysis 1: Comparison: ION-ASD vs Facilitated Play; Ho=No significant interaction of Group*Time; Test type: Superiority; p = 0.310, Mixed Models Analysis — p-value reported for Group*Time, primary comparison in linear mixed effects model (SRS=Group+Time+Group*Time+VIQ+ γ + ε; VIQ, verbal IQ significant covariate), not adjusted for multiple tests (with different time points); Beta Coefficient = -.15

17. Secondary Outcome: Rate of Change From Baseline in Social Functioning (SRS-2)
Description: as for outcome 16
Time Frame: Baseline and Week 12 (Endpoint)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: scores/week
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
scores/week | -.36 (0.21) | -.06 (0.21)

18. Secondary Outcome: Change From Baseline in Social Functioning (SRS-2)
Description: as for outcome 16
Time Frame: Baseline and Week 16 (1-month follow-up)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
T-score
  Estimated mean (baseline) | 70.88 (2.01) | 69.56 (2.07)
  Estimated mean (week 16) | 65.42 (2.01) | 68.69 (2.11)
Statistical Analysis 1: Comparison: ION-ASD vs Facilitated Play; Ho=No significant interaction of Group*Time; Test type: Superiority; p = 0.115, Mixed Models Analysis — [p-value comment as in outcome 16, analysis 1]; Beta Coefficient = -.20

19. Secondary Outcome: Rate of Change From Baseline in Social Functioning (SRS-2)
Description: as for outcome 16
Time Frame: Baseline and Week 16 (1-month follow-up)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: scores/week
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
scores/week | -.34 (0.12) | -0.05 (0.13)

20. Secondary Outcome: Change From Baseline in Social Functioning (SRS-2)
Description: as for outcome 16
Time Frame: Baseline and Week 24 (3-month follow-up)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: T-score
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
T-score
  Estimated mean (baseline) | 69.42 (1.96) | 69.13 (2.00)
  Estimated mean (week 24) | 67.84 (2.05) | 69.74 (2.11)
Statistical Analysis 1: Comparison: ION-ASD vs Facilitated Play; Ho=No significant interaction of Group*Time; Test type: Superiority; p = 0.455, Mixed Models Analysis — [p-value comment as in outcome 16, analysis 1]; Beta Coefficient = -.08

21. Secondary Outcome: Rate of Change From Baseline in Social Functioning (SRS-2)
Description: as for outcome 16
Time Frame: Baseline and Week 24 (3-month follow-up)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: scores/week
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
scores/week | -.07 (0.09) | 0.03 (0.09)

22. Secondary Outcome: Change From Baseline in Quality of Life (CGSQ)
Description: The change from baseline in the Caregiver Strain Questionnaire (CGSQ) is represented by the slope of each group. The primary outcome is the difference between groups in this rate of change or the group*time interaction. The CGSQ was used to assess quality of life. The CGSQ is a parent-rated questionnaire designed for parents of children and adolescents with emotional and behavioral disorders. It includes 21 items rated on a 5-point problem scale (1 = not at all to 5 = very much) rating subjective internal, subjective external, and objective strain. A global measure of strain can be calculated by averaging the scores together. Higher CGSQ scores indicate greater strain. Larger, negative slopes reflect a greater reduction in strain (i.e., improvement in score).
Time Frame: Baseline and Week 12 (Endpoint)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
units on a scale
  Estimated mean (baseline) | 2.52 (0.16) | 2.24 (0.16)
  Estimated mean (week 12) | 2.28 (0.16) | 2.23 (0.16)
Statistical Analysis 1: Comparison: ION-ASD vs Facilitated Play; Ho=No significant interaction of Group*Time; Test type: Superiority; p = 0.379, Mixed Models Analysis — p-value reported for Group*Time, primary comparison in linear mixed effects model (CGS=Group+Time+Group*Time+ γ + ε), not adjusted for multiple tests (with different time points); Beta Coefficient = -.14

23. Secondary Outcome: Rate of Change From Baseline in Quality of Life (CGSQ)
Description: as for outcome 22
Time Frame: Baseline and Week 12 (Endpoint)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: units on a scale/week
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
units on a scale/week | -0.02 (0.02) | 0.00 (0.02)

24. Secondary Outcome: Change From Baseline in Quality of Life (CGSQ)
Description: as for outcome 22
Time Frame: Baseline and Week 16 (1-month follow-up)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
units on a scale
  Estimated mean (baseline) | 2.52 (0.15) | 2.25 (0.15)
  Estimated mean (week 16) | 2.19 (0.15) | 2.15 (0.15)
Statistical Analysis 1: Comparison: ION-ASD vs Facilitated Play; Ho=No significant interaction of Group*Time; Test type: Superiority; p = 0.275, Mixed Models Analysis — [p-value comment as in outcome 22, analysis 1]; Beta Coefficient = -.14

25. Secondary Outcome: Rate of Change From Baseline in Quality of Life (CGSQ)
Description: as for outcome 22
Time Frame: Baseline and Week 16 (1-month follow-up)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: units on a scale/week
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
units on a scale/week | -0.02 (0.01) | -0.01 (0.01)

26. Secondary Outcome: Change From Baseline in Quality of Life (CGSQ)
Description: as for outcome 22
Time Frame: Baseline and Week 24 (3-month follow-up)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
units on a scale
  Estimated mean (baseline) | 2.50 (0.15) | 2.22 (0.15)
  Estimated mean (week 24) | 2.11 (0.16) | 2.22 (0.16)
Statistical Analysis 1: Comparison: ION-ASD vs Facilitated Play; Test type: Superiority; p = 0.087, Mixed Models Analysis — [p-value comment as in outcome 22, analysis 1]; Beta Coefficient = -.20

27. Secondary Outcome: Rate of Change From Baseline in Quality of Life (CGSQ)
Description: as for outcome 22
Time Frame: Baseline and Week 24 (3-month follow-up)
Population: All participants contributed to the intent to treat (ITT) model.
Measure: Mean (Standard Error); unit: units on a scale/week
Arm/Group | ION-ASD | Facilitated Play
Number analyzed (Participants) | 20 | 20
units on a scale/week | -0.02 (0.01) | 0.00 (0.01)

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Systematic assessment of adverse events (AEs) occurred via trained clinician administration of a safety questionnaire (Adverse Event Form) to caregivers typically every other week beginning at week 1. AEs reported by caregivers' calls outside these visits were recorded as non-systematic. Note all severe AEs were for a single participant in the control (Facilitated Play) group. No AEs were rated as related to study drug.
Arm/Group | ION-ASD | Facilitated Play
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 20/20 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ION-ASD (N=20) | Facilitated Play (N=20)
Impulsivity (Psychiatric disorders) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Irritable (Psychiatric disorders) | 0 (0) | 1 (1)
Mood lability (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ION-ASD (N=20) | Facilitated Play (N=20)
Allergic reaction (Immune system disorders) | 2 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 3 (5)
Visual change (Eye disorders) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 5 (7)
Change in appetite (Gastrointestinal disorders) | 7 (10) | 12 (14)
Constipation (Gastrointestinal disorders) | 6 (9) | 5 (6)
Cramping (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 3 (3)
Indigestion (Gastrointestinal disorders) | 1 (1) | 2 (3)
Large and frequent stools (Gastrointestinal disorders) | 1 (1) | 0 (0)
Loose stools (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea/vomitting (Gastrointestinal disorders) | 2 (2) | 4 (5)
Change in sleep (General disorders) | 7 (7) | 8 (13)
Change in speech (General disorders) | 3 (3) | 3 (3)
Fever (Infections and infestations) | 4 (4) | 5 (6)
Infection (Infections and infestations) | 3 (3) | 4 (7)
Loss of tooth (Infections and infestations) | 1 (1) | 1 (1)
Toothache (Infections and infestations) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle ache (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Clumsy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Fatigue (Nervous system disorders) | 3 (4) | 2 (2)
Headache (Nervous system disorders) | 7 (12) | 5 (6)
Hyperactivity/Impulsivity (Psychiatric disorders) | 6 (8) | 9 (11)
Staring episode (Nervous system disorders) | 1 (1) | 0 (0)
Abnormal thoughts (Psychiatric disorders) | 1 (1) | 1 (1)
Aggression (Psychiatric disorders) | 8 (10) | 7 (9)
Anxiety (Psychiatric disorders) | 7 (10) | 10 (14)
Confused (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 4 (6) | 4 (5)
Irritable (Psychiatric disorders) | 16 (24) | 13 (24)
Mood lability (Psychiatric disorders) | 10 (16) | 7 (9)
Poor Concentration (Psychiatric disorders) | 8 (8) | 7 (10)
Nose picking (Psychiatric disorders) | 1 (2) | 0 (0)
Pulling on lip skin (Psychiatric disorders) | 1 (1) | 0 (0)
Repetitive behavior/speech (Psychiatric disorders) | 7 (10) | 8 (15)
Sassy - talking back (Psychiatric disorders) | 1 (1) | 0 (0)
Self-injurious behavior (Psychiatric disorders) | 1 (1) | 3 (3)
Fingernail picking (Psychiatric disorders) | 6 (6) | 9 (11)
Hair pulling (Psychiatric disorders) | 2 (2) | 0 (0)
Skin picking (Psychiatric disorders) | 2 (2) | 3 (3)
Stereotypic movement (Psychiatric disorders) | 2 (2) | 3 (4)
Suicidal thoughts (Psychiatric disorders) | 3 (3) | 0 (0)
Tearful (Psychiatric disorders) | 8 (8) | 1 (1)
Tics (Psychiatric disorders) | 5 (10) | 1 (1)
Enuresis (Renal and urinary disorders) | 2 (2) | 3 (3)
Polydipsia, polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Clearing throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 6 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Runny nose (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 6 (10)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 5 (7)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3)
Eczema (Skin and subcutaneous tissue disorders) | 7 (9) | 4 (6)
Rash (Skin and subcutaneous tissue disorders) | 6 (7) | 4 (6)
Flu (Infections and infestations) | 0 (0) | 1 (1)
Low self esteem (Psychiatric disorders) | 0 (0) | 1 (1)
Odynophagia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Social withdrawal (Social circumstances) | 0 (0) | 1 (1)
Visual change (Eye disorders) | 1 (1) | 0 (0)
Indigestion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Poor concentration (Nervous system disorders) | 1 (1) | 0 (0)
Repetitive behavior/speech (Psychiatric disorders) | 1 (1) | 0 (0)
Stereotypic movement (Psychiatric disorders) | 1 (1) | 0 (0)
Increase in flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Enrollment was slowed down during COVID-19 shut down resulting in the study being under-powered and some groups receiving modified protocols. Apriori secondary analyses of maintenance effects resulted in multiple comparisons tests (i.e., at week 16 and 24) which were not corrected to balance type I/type II errors. Additionally, social cognitive stimuli were not counterbalanced; thus, it's unclear whether social cognitive improvements across groups reflect learning or practice effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/64/NCT02918864/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/64/NCT02918864/SAP_001.pdf
  • Informed Consent Form (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/64/NCT02918864/ICF_002.pdf